CLINICAL TRIAL: NCT01489852
Title: Interest of a Steroid Pre-treatment Prior to IVF Protocol With Ovarian Stimulation by Recombinant FSH and With LH Surge Blockage by Daily GnRH Antagonist
Brief Title: Estrogen Pretreatment Prior to GnRH Antagonist Protocol
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gemer (Other)
Responsible Party: Principal Investigator, Dr CEDRIN-DURNERIN Isabelle, principal investigator, Gemer
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E2PRETREATMENT
Record Dates: First submitted 2011-11-28; First posted 2011-12-12 (Estimated); Last update posted 2011-12-12 (Estimated); Status verified 2011-12

CONDITIONS: Infertility
Keywords: Assisted reproductive treatment; GnRH antagonist; Estrogen pre-treatment; Ovarian stimulation
MeSH Terms: conditions — Infertility | interventions — Estradiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Estrogen pre-treatment (Active Comparator)
  Interventions: Drug: 17beta-estradiol
- Control (No Intervention): The control group did not receive any pre-treatment.

INTERVENTIONS:
Drug: 17beta-estradiol — Pretreatment with 17beta-estradiol (Provames®, Aventis, Paris, France) was administered daily (2 mg twice a day) during the cycle preceding the IVF/ICSI cycle, starting 7 days before the predicted onset of menses and administered up until to the following Thursday after the occurrence of menses.
  Arms: Estrogen pre-treatment

SUMMARY:
The purpose of this study is to assess whether estrogen pre-treatment can allow retrieval of 2 additional oocytes in GnRH antagonist protocol.

ELIGIBILITY:
Inclusion Criteria:

* regular normo-ovulatory cycles (28 to 35 days)
* age < 38 years,
* body mass index (BMI) between 18 and 30
* first or second IVF/ICSI attempt

Exclusion Criteria:

* high basal levels of serum FSH or E2,
* less than 5 follicles at the antral follicular count performed on day 3 of a spontaneous cycle,
* history of high (>20 oocytes) or low (< 5 oocytes) ovarian response in a previous IVF attempt

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 472 (Actual)
Dates: Start 2006-12; Primary Completion 2010-07 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
number of retrieved oocytes | at the ovarian puncture, 36 hours post HCG administration

SECONDARY OUTCOMES:
pregnancy rate | at pregnancy test and at 6 Week US examination
delivery rate | 9 months later
number of obtained embryos | 2 days after in vitro fertilization
duration of FSH administration | at the end of ovarian stimulation usually after a mean of 12 days of administration
  number of days of administration
Total FSH dose | at the end of ovarian stimulation usually after a mean of 12 days of administration
  daily dose x number of days of administration

CONTACTS AND LOCATIONS:
Overall Officials: Jean Noel Hugues, MD, PhD, Study Director — Hôpital Jean Verdier; Isabelle cedrin-durnerin, MD, Principal Investigator — Hôpital Jean Verdier
Locations (1):
- Service de Medecine de la Reproduction, Hôpital Jean Verdier, Bondy, Île-de-France Region, France

REFERENCES:
- [Derived] Cedrin-Durnerin I, Guivarc'h-Leveque A, Hugues JN; Groupe d'Etude en Medecine et Endocrinologie de la Reproduction. Pretreatment with estrogen does not affect IVF-ICSI cycle outcome compared with no pretreatment in GnRH antagonist protocol: a prospective randomized trial. Fertil Steril. 2012 Jun;97(6):1359-64.e1. doi: 10.1016/j.fertnstert.2012.02.028. Epub 2012 Mar 28. PMID 22464760